CLINICAL TRIAL: NCT07121465
Title: The Effect of a Breastfeeding and Infant Care Education Program Prepared According to Mercer Theory on Breastfeeding Self-Efficacy, Readiness for Infant Care, and Acceptance of the Maternal Role
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Antalya Bilim University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ABU-007
Record Dates: First submitted 2025-07-29; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Pregnancy; Breastfeeding; Infant Care; Newborn Care; Theory; Maternal Health
MeSH Terms: conditions — Breast Feeding | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education group (Experimental): First stage: Pregnant women will be administered a "Personal Information Form," the "Prenatal Breastfeeding-Self-Efficacy Scale," the "Prenatal Hygiene Care Readiness Scale," and the "Prenatal Self-Assessment Scale-Maternal Role Acceptance Subscale." Second stage: In this stage, pregnant women will be given a 60-minute breastfeeding education session.
  Third stage: This stage will take place one week after the second stage, and pregnant women will receive baby care training. The training will be conducted face-to-face in the training room of the hospital where the study will be conducted, using the training manual prepared by the researchers according to Mercer's theory as a guide.
  Fourth stage: In this stage, pregnant women will again be administered the "Prenatal Breastfeeding-Self-Efficacy Scale," the "Prenatal Hygiene Care Readiness Scale," and the "Prenatal Self-Assessment Scale-Maternal Role Acceptance Subscale."
  Interventions: Behavioral: Education group; Behavioral: Control group
- Control group (No Intervention): Pregnant women who have not received training will be included in this group.

INTERVENTIONS:
Behavioral: Education group — First stage: Pregnant women will be administered a "Personal Information Form," the "Prenatal Breastfeeding-Self-Efficacy Scale," the "Prenatal Hygiene Care Readiness Scale," and the "Prenatal Self-Assessment Scale-Maternal Role Acceptance Subscale." Second stage: In this stage, pregnant women will be given a 60-minute breastfeeding education session.
  Third stage: This stage will take place one week after the second stage, and pregnant women will receive baby care training. The training will be conducted face-to-face in the training room of the hospital where the study will be conducted, using the training manual prepared by the researchers according to Mercer's theory as a guide.
  Fourth stage: In this stage, pregnant women will again be administered the "Prenatal Breastfeeding-Self-Efficacy Scale," the "Prenatal Hygiene Care Readiness Scale," and the "Prenatal Self-Assessment Scale-Maternal Role Acceptance Subscale."
  Arms: Education group
Behavioral: Control group — First stage: In this stage, pregnant women will be informed about the study and their voluntary written consent will be obtained. They will then complete a Personal Information Form, the Prenatal Breastfeeding Self-Efficacy Scale, the Prenatal Hygienic Care Readiness Scale, and the Prenatal Self-Assessment Scale-Maternal Role Acceptance Subscale.
  Second stage: Pregnant women will be administered the Prenatal Breastfeeding Self-Efficacy Scale, the Prenatal Hygienic Care Readiness Scale, and the Prenatal Self-Assessment Scale-Maternal Role Acceptance Subscale.
  Arms: Education group

SUMMARY:
This study aims to examine the effects of a breastfeeding and infant care education program, developed based on Mercer's Maternal Role Development Theory, on pregnant women's breastfeeding self-efficacy, readiness for infant care, and acceptance of the maternal role. The randomized controlled trial will be conducted with 142 pregnant women between 28 and 32 weeks of gestation who have not received any prior structured education. Data will be collected using the "Personal Information Form," the "Prenatal Breastfeeding-Self-Efficacy Scale," the "Pregnant Women's Readiness for Newborn Hygienic Care Scale," and the "Prenatal Self-Assessment Scale-Maternal Role Acceptance Subscale." Pregnant women in the experimental group will receive a two-session face-to-face education program (breastfeeding and infant care) based on Mercer's theory. One week after the training, participants will be asked to complete the same scales again. Project management included determining the sample size using G*Power, conducting randomization, and analyzing the data using SPSS. The research will be conducted with ethics committee approval, and participant rights will be strictly adhered to.

The broad impact of this study is that structured prenatal education can improve mothers' breastfeeding success and readiness for infant care, facilitating the transition to the motherhood role. The project, which aims to fill gaps in the literature, will contribute to both midwifery practice and evidence-based contributions to maternal and infant health.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who volunteered to participate in the study were:
* 18-35 years old,
* Primiparous,
* Able to speak and understand Turkish,
* 28-32 weeks pregnant,
* Singleton pregnant,
* Having not received any structured education during pregnancy.

Exclusion Criteria:

* Pregnant women with diagnosed mental health problems,
* Those with high-risk pregnancies,
* Those with communication problems,
* Those who do not wish to participate in the study.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 142 (Actual)
Dates: Start 2025-05-30 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-12-28 (Estimated)

PRIMARY OUTCOMES:
Pregnant Women's Readiness Scale for Newborn Hygienic Care | It was applied before and 1 week after the training.
  The scale was developed by Çaka and Çınar in 2020 and consists of 10 items. The scale is a 7-point Likert-type scale, and each item is scored between 1 and 7, from "I'm not ready" to "I'm completely ready." The total scale score is obtained by summing the scores. The minimum score is 10 and the maximum score is 70. High scores indicate a high level of readiness for the pregnant woman. While the validity and reliability of the scale was conducted in primigravida pregnant women, it can also be used in multigravida pregnant women from the second trimester until birth. Scale score evaluation is as follows; 1-3 points: Not ready for hygienic care of the newborn, 4-5: Moderate readiness for hygienic care of the newborn, 6 and above: Readiness for hygienic care of the newborn. The Chronbach's Alpha value of the scale is 0.93 (Çaka et al., 2020).
Prenatal Breastfeeding-Self-Efficacy Scale | It was applied before and 1 week after the training.
  It was developed by Wells et al. in 2006 to determine the perception of breastfeeding self-efficacy in pregnant women during the prenatal period (Wells et al., 2006). The validity and reliability of the Turkish version were conducted by Aydın and Pasinlioğlu. The Cronbach's Alpha value of the scale is 0.86. The scale consists of a total of 20 items. Each item of the scale is rated on a 5-point Likert-type scale: "1 = Not at all sure," "2 = Somewhat sure," 3 = Fairly sure," 4 = Very sure," and 5 = Absolutely sure." It has no sub-dimensions. It is evaluated based on a total score. The lowest score that can be obtained from the total scale is 20, and the highest score is 100. A higher score indicates an increase in the perception of breastfeeding self-efficacy (Aydın & Pasinlioğlu, 2018).
Prenatal Self-Assessment Scale-Maternal Role Acceptance Subscale | It was applied before and 1 week after the training.
  Developed by Lederman in 1979, it is a measurement tool used to assess pregnant women's adjustment to pregnancy and motherhood. The scale's validity and reliability study in Turkey was conducted by Beydağ and Mete (2008). The scale contains 7 subscales and 79 items. The internal consistency coefficient of the scale translated into Turkish was found to be Cronbach's alpha 0.81, and the internal consistency reliability coefficients of the subgroups ranged from 0.72 to 0.85 (Beydağ and Mete 2008). The 15-item Acceptance of the Motherhood Role subscale will be used in the study. Adjustment to pregnancy is assessed based on scores ranging from 1 to 4 (4: Very much describes, 3: Partially describes, 2: Somewhat describes, 1: Not at all describes). Scoring is reversed for reversed items. The lowest possible score from the maternal role acceptance subscale is 15, and the highest is 60. A low score indicates high compliance (Beydağ & Mete, 2008).

CONTACTS AND LOCATIONS:
Locations (1):
- Antalya Bilim Üniversitesi, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The study will be shared after it is published.